CLINICAL TRIAL: NCT01346176
Title: The Influence of Default Options in Advance Directives for Older Patients: A Pilot Study
Brief Title: The Influence of Default Options in Advance Directives
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Scott Halpern, Assistant Professor of Medicine, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 810894
Record Dates: First submitted 2011-04-29; First posted 2011-05-02 (Estimated); Results first posted 2016-02-03 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-01

CONDITIONS: Advance Care Planning

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Positive default (Experimental): Patients in this arm will receive AD forms where specific life-extending interventions will be provided unless patients specifically opt-out from such selections
  Interventions: Other: Advance Directive Forms
- Negative default (Experimental): Patients in this arm will receive AD forms where specific life-extending interventions will not be provided unless patients specifically opt-into such selections
  Interventions: Other: Advance Directive Forms
- Forced Choice (Experimental): Patients in this arm will receive AD forms in which they must actively choose whether to receive each intervention.
  Interventions: Other: Advance Directive Forms

INTERVENTIONS:
Other: Advance Directive Forms — Consenting subjects will be randomly assigned to one of 3 study arms. Subjects will receive a different AD form based on which arm they have been randomly assigned. Once a completed AD form is received, a debriefing session will be held to alert patients to exactly how the 3 ADs used in the study differ. Once patients are fully informed about the variations in the ADs, they will have an opportunity to change their AD selections prior to finalizing them as a part of their medical record. A final satisfaction interview will take place with a research associate who will contact patients via telephone to administer a satisfaction questionnaire.

SUMMARY:
The investigators aim to assess the influence of default options in advance directives on older patients selections of life- extending therapies and to determine whether alerting patients to the spectrum of possible default options in advance directives influences their selections of life-extending therapies by manipulating the default options of advance directives given to patients in with severe respiratory disease

DETAILED DESCRIPTION:
The project is designed to document that default options influence terminally ill patients end-of-life decisions (in this case, adults with advance forms of lung disease) and that our team can recruit and retain patients in a study of advance care planning. In addition, because a larger-scale randomized clinical trial will require that the investigators alert participants to the range of possible default options, the investigators must also determine the effects that this alerting will have on their selections of life-extending therapies. Therefore, the investigators seek to achieve three aims: (1) assess the influence of default options in advance directives on patients selections of life-extending therapies; (2) determine whether alerting patients to the spectrum of possible default options in advance directives influences their selections of life extending therapies; and (3) document the feasibility of recruiting and retaining patients with advanced lung diseases from university-based clinical settings into a randomized trial of default options in advance directives.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic obstructive pulmonary disease (COPD), idiopathic pulmonary fibrosis (IPF), non-small-cell lung cancer, or other interstitial or fibrotic lung disease
* Neither listed for nor considering solid organ transplantation
* Anticipated survival of less than 2 years
* Must be fluent and literate in English

Exclusion Criteria:

* Diagnosis of small-cell lung cancer or other respiratory diseases for which life extending medical therapies may be available

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2010-04; Primary Completion 2012-03 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott D. Halpern, MD, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania School of Medicine, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place in outpatient clinics at the Pereleman Center for Advanced Medicine at the University of Pennsylvania. Recruitment occurred from May 2010 - Feb 2012. No recruitment occurred between Oct 2010 - Jan 2011 while the first research nurse transitioned responsibilities to the second research nurse.
Pre-assignment Details: 9,378 patients were assessed for eligibility. 9,246 were excluded. 8,299 did not meet inclusion criteria, 391 already had an advance directive, 322 were either missed in clinic, cancelled their appointments, or were hospitalized, 181 declined participation, 43 had their participation deferred by their physician
Period: Recruited
Arm/Group | Positive Default | Negative Default | Forced Choice
Started | 49 | 40 | 43
Completed | 48 | 40 | 43
Not Completed | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Period: Completed Advance Directive
Arm/Group | Positive Default | Negative Default | Forced Choice
Started | 48 | 40 | 43
Completed | 35 | 26 | 33
Not Completed | 13 | 14 | 10
Not completed — Death | 3 | 2 | 2
Not completed — Became Ineligible | 3 | 0 | 1
Not completed — Other reason did not complete AD | 7 | 12 | 7
Period: Completed Satisfaction Survey
Arm/Group | Positive Default | Negative Default | Forced Choice
Started | 35 | 26 | 33
Completed | 29 | 22 | 27
Not Completed | 6 | 4 | 6
Not completed — Death | 3 | 0 | 2
Not completed — Lost to Follow-up | 3 | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Positive Default | Negative Default | Forced Choice | Total
Number analyzed (Participants) | 49 | 40 | 43 | 132
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.6 (8.50) | 64.8 (8.61) | 64.4 (7.12) | 64.63 (8.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 23 | 28 | 76
  Male | 24 | 17 | 15 | 56
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 11 | 10 | 14 | 35
  White | 34 | 28 | 29 | 91
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 4 | 2 | 0 | 6

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Who Select Palliative Care Options
Description: The primary outcome variable will be the proportion of subjects that select palliative care options compared to the those who request aggressive treatment in each study arm. We will analyze the effects of manipulating default options and delays in alerting subjects to the presence of multiple default options on each selection in the ADs in order to see how default options influence decisions on general treatment goals and instructions for specific procedures.
Time Frame: 6 months
Population: This number was based on the number of participants who returned completed advance directive forms in each group
Measure: Number (95% Confidence Interval); unit: percentage who select palliative care
Arm/Group | Positive Default | Negative Default | Forced Choice
Number analyzed (Participants) | 48 | 40 | 43
percentage who select palliative care | 31 [19 to 46] | 50 [34 to 66] | 47 [31 to 62]

2. Secondary Outcome: Patient Satisfaction With Advance Care Planning.
Description: Patients' satisfaction with their advance care planning was assessed two months after they completed their ADs. One of two authors blinded to patients' group assignments contacted patients by phone and administered a satisfaction survey based on the Canadian Healthcare Evaluation Project (CANHELP) questionnaire. This thirteen-item questionnaire has been validated for assessing satisfaction with end-of-life care planning. Patients were asked to indicate satisfaction with various parts of advance care planning (e.g. decisions about the use of life sustaining technologies including CPR or cardiopulmonary resuscitation, breathing machines, and dialysis) on a scale from 1 to 5, where 1 means not at all satisfied and 5 means completely satisfied. The overall average across the 13 item scale in each group is presented in the results below.
Time Frame: Two months after AD completion
Population: These numbers reflect the number of patients who completed and returned and advance directive as well as completed a satisfaction interview and questionnaire with a research associate.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Positive Default | Negative Default | Forced Choice
Number analyzed (Participants) | 29 | 22 | 27
units on a scale | 4.51 [1 to 5] | 4.61 [1 to 5] | 4.56 [1 to 5]

ADVERSE EVENTS:
Arm/Group | Forced Choice | Negative Default | Positive Default
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/49 | 0/40 | 0/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Forced Choice (N=0) | Negative Default (N=0) | Positive Default (N=0)
Serious adverse events not reported (Investigations) | 0 (0) | 0 (0) | 0 (0) — This was a minimal risk study, patients were not at risk for any serious adverse events. Serious adverse events were not collected or reported.

LIMITATIONS AND CAVEATS:
1. This is a small sample from a single health system
2. Limited to patients with serious thoracic diseases
3. We did not randomly assign the ordering of options within the standard advance directive

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No